CLINICAL TRIAL: NCT07334756
Title: Non-Thrust Lumbar and Sacral Mobilizations in Mechanical Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/27
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded about the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: lumbar mobilization (Active Comparator): Lumbar mobilizations along with the standard therapeutic exercise protocol.
  Interventions: Procedure: Lumbar Mobilizations
- Group B: Sacral mobilizations+lumbar mobilization (Experimental): Sacral mobilizations in addition to the lumbar mobilization and therapeutic exercise.
  Interventions: Procedure: Lumbar and sacral mobilizations

INTERVENTIONS:
Procedure: Lumbar Mobilizations — Lumbar mobilization protocol:
  Grade II or III lumbar stretch mobilization on lumbar hypomobile segments.
  Therapeutic exercise protocol:
  Therapeutic exercise protocol include warmup, strengthening and cool down phase.
  Arms: Group A: lumbar mobilization
Procedure: Lumbar and sacral mobilizations — Lumbar mobilization protocol:
  Grade II or III lumbar stretch mobilization on lumbar hypomobile segments.
  Sacral Mobilization protocol:
  Grade II or III sacral mobilization as sacral stretch mobilizations.
  Therapeutic exercise protocol:
  Therapeutic exercise protocol include warmup, strengthening and cool down phase.
  Arms: Group B: Sacral mobilizations+lumbar mobilization

SUMMARY:
This study is a randomized controlled trial and the purpose of this study is to determined the effects of sacral mobilizations along with the lumbar mobilizations in mechanical low back pain on components such as pain , lumbar range of motion, lumbar proprioception and functional disability.

DETAILED DESCRIPTION:
This study is based on the concept the sacral hypomobility can cause low back pain. Sacral and lumbar mobilizations both improve low back pain.

ELIGIBILITY:
* Inclusion Criteria Adults 18 to 45 years Both genders Low back (from T12 to buttock line) pain for more than 3 months The CMLBP is the chief complaint without leg pain.
* Exclusion Criteria Acute flare Low Back Pain Thoracic pain Trauma to the spine causing fracture and disruption of the ligaments Leg symptoms when walk, eased in flexion (Signs of stenosis) Paresthesia/numbness Structural deformity (scoliosis, spondylosis, spondylolisthesis) Curve reversal Pregnancy Post-surgery (within 6 months of abdominal or spinal/lower limb surgery) Degenerative and inflammatory spinal diseases Malignancy Centralization and peripheralization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Numeric pain scale rating (NPRS) w3ill be used and It ranges from 0 to 10, 0 means no pain and 10 means worst pain.
Lumbar Range of Motion | 2 weeks
  It will be measured by Inclinometer . it is Measured by placing the inclinometers at T12 and S1.
Functional Disability | 2 weeks
  It will be measured by Oswestry Disability Index. It is a 10 items questionnaire used to assess the degree of disability in individuals with low back pain.
Lumbar Proprioception | 2 weeks
  it is measured by Joint position sense/ error test . it is Measured by placing the inclinometers at T12 and S1.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Punjab Province, Pakistan